CLINICAL TRIAL: NCT00738933
Title: Effects of Dietary Plant Sterols and Stanols on Sterol Composition and Structure of the Human Aortic Valve
Brief Title: Dietary Phytosterols and Human Aortic Valve
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Helsinki (Other)
Collaborators: University of Eastern Finland (Other)
Responsible Party: Markku Nissinen, MD PhD, Helsinki University Central Hospital
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 231857
Record Dates: First submitted 2008-08-20; First posted 2008-08-21 (Estimated); Last update posted 2011-02-14 (Estimated); Status verified 2011-02

CONDITIONS: Hypercholesterolemia; Atherosclerosis
Keywords: Atherosclerosis; Plant sterols; Plant stanols; Aortic valve
MeSH Terms: conditions — Hypercholesterolemia; Atherosclerosis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- A (Active Comparator): A group of patients consuming 2 grams plant stanols 4-8 weeks before the operation
  Interventions: Dietary Supplement: Dietary plant stanols
- E (Active Comparator): A group of patients consuming daily 2 grams plant sterols 4-8 weeks before the operation.
  Interventions: Dietary Supplement: Dietary plant sterols
- C (Placebo Comparator)
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: Dietary plant stanols — Daily 2 grams of plant stanols in a margarine preparation for 4-8 weeks before the operation
  Arms: A
Dietary Supplement: Dietary plant sterols — Daily 2 grams of plant sterols in a margarine preparation for 4-8 weeks before the operation
  Arms: E
Dietary Supplement: placebo — Margarine product without plant stanol or sterol esters
  Arms: C

SUMMARY:
This randomized controlled double-blind intervention study unravels influence of dietary plant sterols and stanols on the structure and the sterol composition of the human aortic valve. The study patients will include 50-60 voluntary patients from the Helsinki Univ. Central Hospital, who will undergo aortic valve surgery. The patients will be randomized into plant sterol (E), plant stanol (A) and control (C) groups. Patients in the E and A groups will be asked to consume daily 2 grams plant sterols or plant stanols, respectively, in a margarine product.

DETAILED DESCRIPTION:
High level of serum cholesterol is a risk factor for atherosclerotic complications, including atherosclerotic aortic valve disease. Over 50 years dietary plant sterols have been used to inhibit intestinal cholesterol absorption and to decrease its levels in serum. Daily human diet contains numerous different plant sterols, of which sitosterol and campesterol are the most abundant ones. Few epidemiologic studies suggest that sitosterol and campesterol may also be involved in formation of atherosclerotic changes in human arteries. The saturated forms of sitosterol and campesterol, i.e., the plant stanols (mainly sitostanol and campestanol) are beneficial with this respect. As part of daily diet, the plant stanols decrease absorption of both cholesterol and plant sterols, and thus, are putatively even more effective in prevention of atherosclerosis than the respective plant sterols.

Our double-blind controlled intervention study unravels influence of dietary plant sterols and stanols on the structure and the sterol composition of the human aortic valve.

50-60 patients, who will undergo aortic valve surgery, will be asked to volunteer our study. The patients will be randomized into three groups: (A) a group consuming margarine containing daily 2 grams plant stanols, (E) a group consuming margarine containing daily 2 grams of plant sterols, (C) a control group consuming margarine without any plant sterols or stanols. The dietary intervention will last for 4 to 8 weeks from the randomization to the operation.

Serum samples for analyses of serum lipids, lipoproteins and sterols will be collected at the randomization and at the operation. The atherosclerotic aortic valve will be examined with respect to its composition of cholesterol, other sterols and stanols.

The aim of our study is to elucidate the effects of dietary consumption of plant sterols and stanols on the sterol composition and structure of the atherosclerotic disease-affected aortic valve in human patients.

ELIGIBILITY:
Inclusion Criteria:

* Atherosclerotic aortic valve disease needing an aortic valve replacement operation

Exclusion Criteria:

* None

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2008-04; Primary Completion 2011-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Composition of serum and aortic valve sterols at the time of aortic valve operation | Up to 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Tatu A. Miettinen, professor, Principal Investigator — Dept. of Medicine, Div. of Internal Medicine, Helsinki Univ. Central Hospital, Biomedicum Helsinki; Helena Gylling, Professor, Principal Investigator — Department of Clinical Nutrition, University of Kuopio and Kuopion University Central Hospital, Kuopio, Finland; Markku J Nissinen, MD, PhD, Principal Investigator — Dept. of Medicine, Div. of Gastroenterology, HUCH, Helsinki, Finland
Locations (1):
- Department of Medicine, Div. of Internal Medicine, Helsinki Univ. Central Hospital (HUCH), Helsinki, Finland

REFERENCES:
- [Derived] Simonen P, Stenman UH, Gylling H. Serum proprotein convertase subtilisin/kexin type 9 concentration is not increased by plant stanol ester consumption in normo- to moderately hypercholesterolaemic non-obese subjects. The BLOOD FLOW intervention study. Clin Sci (Lond). 2015 Sep;129(5):439-46. doi: 10.1042/CS20150193. Epub 2015 Apr 10. PMID 25857271
- [Derived] Simonen P, Lommi J, Hallikainen M, Helske-Suihko S, Werkkala K, Kupari M, Kovanen PT, Gylling H. Dietary plant stanols or sterols neither accumulate in stenotic aortic valves nor influence their structure or inflammatory status. Clin Nutr. 2015 Dec;34(6):1251-7. doi: 10.1016/j.clnu.2015.01.001. Epub 2015 Jan 7. PMID 25614126